CLINICAL TRIAL: NCT01533896
Title: Can a Brief Primary Care Intervention Affect Healthy Weight Habits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Seth Scholer, Associate Professor of Pediatrics, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: grownicely
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Obesity
Keywords: Obesity prevention; Primary care; Education
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Parents and children in the control group received routine primary care during the well child visit.
- Grow Nicely (Experimental): Grow Nicely multimedia program.
  Interventions: Behavioral: Grow Nicely

INTERVENTIONS:
Behavioral: Grow Nicely — Grow Nicely is a multimedia educational tool, developed at Vanderbilt University that teaches why and how to help children reach and maintain a healthy weight.
  Arms: Grow Nicely

SUMMARY:
Parents should receive anticipatory guidance about obesity prevention as part of the routine well child visit. Educational resources are needed to help physicians routinely provide these important anticipatory guidance messages. In this study, consecutive parents will be exposed to routine anticipatory guidance messages before the well child visit with the physician. After the clinic visit, parents will be invited to participate in a research study to determine if they plan any changes at home. The key research question of this study is: Can a brief multimedia intervention help parents develop plans to help their children have a healthy weight?

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speaking parents of 2-12 year old children presenting to the pediatric primary care clinic.

Exclusion Criteria:

* Parent does not speak English or Spanish.
* Child presenting for an acute care visit.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Changes in healthy weight habits | 2 -4 weeks
  At the time of the follow up phone call 2-4 weeks post-intervention, parents were asked: "Since the clinic visit have you made any changes to help your child either reach or maintain a healthy weight? "
  * Yes "If yes, what changes have you made?"

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Pediatric Primary Care Clinic, Nashville, Tennessee, United States